CLINICAL TRIAL: NCT00873756
Title: A Phase Ib Study of the Safety and Pharmacokinetics of Dulanermin Administered in Combination With the FOLFOX Regimen and Bevacizumab in Patients With Previously Untreated, Locally Advanced, Recurrent, or Metastatic Colorectal Cancer
Brief Title: A Study of Dulanermin Administered in Combination With the FOLFOX Regimen and Bevacizumab in Patients With Previously Untreated, Locally Advanced, Recurrent, or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APO4565g; GO00934 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-03-05; First posted 2009-04-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: CRC; Colon Cancer; Avastin; Apo2L/TRAIL
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Folfox protocol; Bevacizumab; TNFSF10 protein, human

ARMS (1):
- A (Experimental)
  Interventions: Drug: FOLFOX regimen; Drug: bevacizumab; Drug: dulanermin

INTERVENTIONS:
Drug: FOLFOX regimen — Intravenous repeating dose
Drug: bevacizumab — Intravenous repeating dose
Drug: dulanermin — Intravenous repeating dose

SUMMARY:
This is a multicenter, open-label study enrolling a total of up to 23 patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CRC with evidence of locally advanced recurrent or metastatic disease (i.e., by radiographic imaging or biopsy) and measurable tumor lesions
* Life expectancy > 3 months
* For patients of reproductive potential (males and females), use of reliable means for contraception throughout the trial
* Willingness and capability to be accessible for study follow-up

Exclusion Criteria:

* Prior 5-FU, capecitabine, and/or oxaliplatin treatment with the exception of: prior oxaliplatin treatment =< 6 weeks in the advanced or metastatic setting; prior treatment with 5-FU, capecitabine, and/or oxaliplatin in the adjuvant setting if relapse occurred > 6 months from concluding adjuvant therapy
* Peripheral neuropathy Grade >= 2
* Prior radiotherapy to a measurable metastatic lesion(s) to be used for response assessment, unless the lesion has progressed subsequent to the radiotherapy
* Radiotherapy to a peripheral lesion within 14 days prior to Cycle 1, Day 1, or radiotherapy to a thoracic, abdominal, or pelvic field within 28 days prior to Cycle 1, Day 1
* Chemotherapy, hormonal therapy, or immunotherapy within 4 weeks prior to Cycle 1, Day 1
* Evidence of clinically detectable ascites
* Other invasive malignancies within 5 years prior to Cycle 1, Day 1
* Current or recent participation in another experimental drug study
* Clinically significant cardiovascular disease, New York Heart Association (NYHA) Grade II or greater congestive heart failure, serious cardiac arrhythmia within 1 year prior to Cycle 1, Day 1, or Grade II or greater peripheral vascular disease on Cycle 1, Day 1
* Active infection requiring parenteral antibiotics
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Cycle 1, Day 1, fine needle aspirations or minor surgery (such as port placement) within 7 days prior to Cycle 1, Day 1, or anticipation of need for major surgical procedure during the course of the study
* Known or suspected to be positive for the human immunodeficiency virus (HIV)
* Known to be positive for hepatitis C or hepatitis B surface antigen
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or specified study treatment, or that might affect interpretation of the results of the study or render the patient at high risk from treatment complications
* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History of arterial thromboembolic event 6 months prior to Cycle 1, Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Cycle 1, Day 1
* Bleeding diathesis or coagulopathy
* Pregnancy (positive pregnancy test) or breast feeding
* Serious, non-healing wound, ulcer, or bone fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-05; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities | Until study discontinuation or the end of Cycle 26

SECONDARY OUTCOMES:
Incidence, nature, and severity of adverse events | Until study discontinuation or the end of Cycle 26
Change in vital signs | Until study discontinuation or the end of Cycle 26
Change in clinical laboratory results | Until study discontinuation or the end of Cycle 26
Incidence of anti-dulanermin antibodies | Until study discontinuation or the end of Cycle 26

CONTACTS AND LOCATIONS:
Overall Officials: Chia Portera, M.D., Study Director — Genentech, Inc.
Locations (7):
- United States (7):
  - Los Angeles, California
  - San Francisco, California
  - Aurora, Colorado
  - Fort Collins, Colorado
  - Harvey, Illinois
  - Albuquerque, New Mexico
  - Chapel Hill, North Carolina